CLINICAL TRIAL: NCT04666493
Title: Adapting Anxiety Intervention for Youth With Autism for Rapid Response to COVID-19: A Research Project to Provide and Evaluate Virtual Mental Health Care
Brief Title: Adapting Anxiety Intervention for Youth With Autism for Rapid Response to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0240
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This is a 12 week, single site, single group, open-label trial of the Facing Your Fears intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Facing Your Fears - Open label (Experimental): All participants in the study will receive 12 weekly sessions of Facing Your Fears intervention, each lasting approximately 1 to 1.5 hour. Each session involves a component with all the parents and children (30-45 minutes) and a separate time with all the parents only (30-45 minutes). Additionally, there will be two check-in calls (30 minutes each) with the families after weeks 7 and 9 of the program.
  Interventions: Other: Cognitive behavior therapy (CBT), specifically using the Facing Your Fears (FYF) curriculum

INTERVENTIONS:
Other: Cognitive behavior therapy (CBT), specifically using the Facing Your Fears (FYF) curriculum — The Facing Your Fears program (FYF; Reaven et al. 2011) is a CBT-based group treatment program that has been adapted for the needs of children with high-functioning ASD. The current project will adapt the FYF program for virtual delivery and examine its effectiveness.
  Other Names: Facing Your Fears (FYF)

SUMMARY:
This study will examine if a virtual delivery of a group Cognitive Behavioural Therapy (CBT) program, specifically using "Facing Your Fears" (FYF) curriculum, is helpful in improving anxiety symptoms for children and youth with ASD. This study will adapt the FYF program for virtual delivery using a platform called "Zoom for Healthcare" and examine its effectiveness.

DETAILED DESCRIPTION:
The research team will adapt the Facing Your Fears (FYF) program, in consultation with program developers, Canadian experts (psychologists) and Holland Bloorview's Research Family Engagement Committee, to allow for virtual delivery of a traditionally in-person intervention. Adaptations will build on preliminary work already piloted by program developers to meet the current needs (e.g., group work with individual support, video practice for exposures, psychoeducation format).

Participants will complete one screening phone call and one videoconferencing (Zoom for Healthcare) call with the research team, where the delegated research staff will introduce the program and obtain consent for interested and eligible participants. Participants will be asked to provide consent, then proceed to the second part of the screening to ensure that potential participants meet all eligibility criteria. It will be made clear to participants that providing consent and assent at this time will not guarantee study enrollment.

Once eligibility is confirmed, participants will be enrolled in the study and be asked to provide the study team with the participant's ASD diagnostic letter via a secure link (using Sync), complete pre-intervention questionnaires before the start of the program, and post-intervention questionnaires after completing the study intervention.

The program will be abbreviated from 14 weeks to 12 weeks to maximize the number of families served during the study period. Each session will be approximately 60-90 minutes (30-45 minutes with parents and children; 30-45 minutes with parents alone). There will be two check-in calls (approximately 30 mins) with each of the families after weeks 7 and 9 of the program. The group facilitators will use the Zoom for Healthcare platform to deliver the intervention virtually.

ELIGIBILITY:
Inclusion Criteria:

1. Chronological age between 8 and 13 years (13 yr, 11 mos, 29 days)
2. Have a clinical diagnosis of Autism Spectrum Disorder (ASD)
3. Ability to read at a grade 2 level or above (based on parent report)
4. Verbally fluent at a grade 2 level or above (can speak or respond to questions that are appropriate for a child in grade 2; based on parent report)
5. Child with significant anxiety symptoms as determined by the clinical team
6. To enhance generalizability of our findings, children will be eligible if they present with some other co-morbid psychiatric conditions (see exclusion criteria)
7. If already receiving pharmacological interventions, must meet the following criteria: If receiving concomitant medications for anxiety, must be on a stable dose during the month prior to screening (6 weeks for fluoxetine).

Exclusion Criteria:

1. Being currently enrolled in another active behavioral/ educational/ psychological treatment for anxiety
2. Diagnosis of acute psychosis or conduct disorder, or a primary diagnosis of Obsessive Compulsive Disorder without another anxiety diagnosis or clinically significant level of anxiety.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Screen for Child Anxiety Related Emotional Disorders (SCARED), Parent version | SCARED, Parent version will be administered at baseline (pre-intervention) and at week 12, (post-intervention) to assess change between two time points.
  The SCARED is a 38-item measure of anxious symptoms, with both child and parent versions. The parent version will be used as a primary outcome measure, administered at pre- and post-intervention.

SECONDARY OUTCOMES:
Screen for Child Anxiety Related Emotional Disorders (SCARED), Child version | SSCARED, Child version will be administered at baseline (pre-intervention) and at week 12, (post-intervention) to assess change between two time points.
  The SCARED is a 38-item measure of anxious symptoms, with both child and parent versions. The child version will be used as a secondary outcome measure, administered at pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, MD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brian J, Solish A, Leef J, Nguyen J, Bickle L, Budovitch R, Chan V, Drouillard B, Drumm E, Genore L, Adams RH, Hermolin R, Klemencic N, Lambert M, Lee K, Lim J, Mak-Fan K, O'Neill M, Price S, Pye M, Selezneva E, Taheri A, Anagnostou E. Virtual delivery of group-based cognitive behavioral therapy for autistic children and youth during the COVID-19 pandemic was acceptable, feasible, and effective. Sci Rep. 2025 Feb 27;15(1):7034. doi: 10.1038/s41598-025-88779-7. PMID 40016235